CLINICAL TRIAL: NCT05087199
Title: COVID-19 Infection in Patients With Chronic Pulmonary Diseases.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Elsayed, Principal Investigator, Sohag University
Other Study IDs: OHRP#:IRB00013006
Record Dates: First submitted 2021-10-20; First posted 2021-10-21 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Chronic Pulmonary Disease
Keywords: COVID-19; Chronic pulmonary disease
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rt-PCR. — Nasopharyngeal swab for Rt-PCR for COVID-19
  Other Names: Ct chest; D-dimer; CRP

SUMMARY:
This study aims to assess the clinical presentation, radiological patterns and outcome of COVID-19 infection in patients with chronic pulmonary disease.

Inter-relationship between the severity of COVID-19 infection and chronic pulmonary diseases.

DETAILED DESCRIPTION:
The COVID-19 pandemic has led to many difficulties with the diagnosis and routine management of chronic pulmonary diseases such as COPD, Bronchial asthma, ILD and Bronchiectasis as well as raising concerns about the management and outcomes for patients with these diseases who develop COVID-19.

Although there is conflicting evidence on whether patients with chronic respiratory diseases are more susceptible to COVID-19, these patients exhibit a more severe presentation and higher mortality compared with those without chronic respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of COVID-19 infection by:

RT-PCR And Chest Computed tomography and laboratoty investigations. Patients with chronic chest disease including (COPD, bronchial asthma, ILD, bronchiectasis).

Exclusion Criteria:

* Those who are diagnosed with viral pneumonia caused by viruses other than COVID-19.

Those who are not confirmed to be COVID-19 with PCR or by radiological and laboratory investigations.

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Community sample with chronic pulmonary diseases
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Effect of COVID-19 on patients with chronic pulmonary diseases | 2 weeks after patient confirmation of infection by COVID-19